CLINICAL TRIAL: NCT00126932
Title: Reduction of Topical Anesthetic Onset Time Using Ultrasound: A Randomized Controlled Trial Prior to Venipuncture in Young Children
Brief Title: Reduction of Topical Anesthetic Onset Time Using Ultrasound
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-003
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Device: SonoPrep

SUMMARY:
Children ages 3-7 who are undergoing blood drawing receive either standard care, topical medicine for numbing (LMX4), or the study intervention which utilizes ultrasound to speed the onset of LMX4 from 30 minutes to 5 minutes. The child's pain with the blood drawing procedure is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-7, requiring venipuncture

Exclusion Criteria:

* Emergent procedure
* Allergy to lidocaine or sodium lauryl sulfate

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70
Dates: Start 2004-10; Study Completion 2004-12

PRIMARY OUTCOMES:
pain associated with venipuncture

SECONDARY OUTCOMES:
safety
skin effects
tolerability

CONTACTS AND LOCATIONS:
Overall Officials: William T. Zempsky, MD, Principal Investigator — CT Children's Medical Center
Locations (1):
- CT Children's Medical Center, Hartford, Connecticut, United States